CLINICAL TRIAL: NCT03981679
Title: Prospective, Non-randomized, Open-label and Multi-center Study With the Establishment of a Clinical-biological Database.
Brief Title: Circulating-free DNA Assessment as a Tool to Predict Colorectal Cancer in Subjects With a Positive Fecal Immunoassay.
Acronym: DEPLR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PROICM 2017-02 DEP
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer
Keywords: colonoscopy; CRC screening; cfDNA; Intplex; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): For all the patients include in the study :
  - Blood samples collected before the colonoscopy In parallel to this biological collection, standardized clinical data will be entered into a database
  Interventions: Other: Biological collection

INTERVENTIONS:
Other: Biological collection — The biological collection will also include samples of blood samples collected before colonoscopy

SUMMARY:
Colorectal cancer (CRC): is one of the most frequent cancers, with almost 42152 new cases estimated in France for 2012. There are 3 levels of risk of developing CRC: moderate, high or very high. At each level of risk, appropriate follow-up recommendations are made. Immunological tests for fecal occult blood tests have emerged in recent years and have rapidly become established as benchmark tests in Europe and then in France (OC Sensor test) as part of mass screening. In the case of a positive immunological test, a diagnostic colonoscopy must be systematically organized in order to characterize the possible recto-colic cause of the digestive bleeding thus observed.

Measurement of the DNA present in the circulating blood (circulating DNA or cfDNA): allowed a significant advance in the personalized management of cancers, as a non-invasive test capable of producing diagnostic, prognostic, theranostic, and of therapeutic follow-up type.

The aim of the work is to measure the cfDNA concentration in subjects undergoing colonoscopy because of a positive immunological fecal test.

DETAILED DESCRIPTION:
Colorectal cancer (CRC): is one of the most frequent cancers, with almost 42152 new cases estimated in France for 2012. The incidence is thus 30 new cases per year per 100 000 inhabitants in France. It is also a significant cause of death, with 10 deaths per year per 100,000 inhabitants. More than 8 patients out of 10 are cured by surgery alone in case of discovery of an early form with a tumor extension limited to the colonic wall and absence of proximal lymph node invasion. Since most of the invasive cancers are preceded by a benign precancerous lesion called adenoma, it is well understood that the detection of these adenomas (and in particular those at high risk of cancerization: adenomas greater than 10 mm or adenomas in severe dysplasia), followed by their endoscopic excision (polypectomy via colonoscopy) can prevent the development of invasive CRC and ultimately improve the survival of the population thus detected. It is precisely the possibility of intervening on this sequence adenomacancer during an asymptomatic phase of the disease that is the basis of the offer of screening for CRC. CRC screening: There are 3 levels of risk of developing CRC: moderate, high or very high. At each level of risk, appropriate follow-up recommendations are made.considered moderate risk of developing CRC, subjects older than 50 years. These patients at risk are also the most numerous. They are the ones who are involved in screening for occult blood in the stool. Two methods of screening were recommended for moderate-risk subjects, left-sided recto-sigmoidoscopy and repeated occult blood tests in the faeces by the Gaiac method. The latter method has rapidly became in Europe a reference method for screening CRC for reasons of cost and access to care. However, it appears to be a method which is not very appreciated by patients (manipulation of several stool samples) and which is not very sensitive, and which may also interact with hemoglobin of animal origin. These disadvantages have led to an interest in other methods of screening occult blood in stools, such as immunological methods. Immunological tests for fecal occult blood tests have emerged in recent years and have rapidly become established as benchmark tests in Europe and then in France (OC Sensor test) as part of mass screening. Briefly, 2 Dutch randomized studies showed that the OC Sensor immunoassay had better screening performance and acceptability than the Gaiac test. Overall, the different studies have shown that immunological tests lead to more CRCs and more advanced neoplasia than the Gaiac test. According to the studies, the positivity rate ranged from 3% to 6% for immunoassays, the positive predictive value of advanced neoplasia was about 45% with OC Sensor, and that of invasive cancer was 7%. Thus, the OC Sensor fecal immunoassay is the reference screening test, as part of the organized screening of subjects at moderate risk of CRC. In the case of a positive immunological test, a diagnostic colonoscopy must be systematically organized in order to characterize the possible recto-colic cause of the digestive bleeding thus observed. The colonoscopy identifies the lesion and the biopsies then performed accurately identify the advanced nature (adenoma> 10 mm or adenoma in severe dysplasia or invasive cancer) or not of the neoplasia. Colonoscopy is a perfectly controlled medical procedure performed under anesthesia.

It can, however, exceptionally cause bleeding, perforation of the colon, severe abdominal pain, especially when the endoscopic act is associated with an interventional act such as biopsy or polypectomy. The practice of colonoscopy is yearly responsible for 3 accidents on 1000 colonoscopies performed, leading to 1 surgery on 1000 colonoscopy, and unfortunately to 1 death every 10 000 colonoscopies. Because the colonoscopy is performed under anesthesia, this forces the patient to absent himself from work for one day, to call on a third party to return home. Finally, although colonoscopy is the most sensitive and specific test for the diagnosis of adenomas and CRCs, its diagnostic performance is not absolute: complete colon exploration is only possible in 95 % Of cases. Colonoscopy is missing in particular 5% of adenomas of more than 1 cm and 4% of colon cancers of the right colon. Colonoscopy also has a cost. Thus, any non-invasive test capable of making a diagnosis of invasive cancer or discarding the same cancer diagnosis after a positive immunological fecal screening test would be able to reduce the use of diagnostic colonoscopy and thus the risks and Associated constraints. Measurement of the DNA present in the circulating blood (circulating DNA or cfDNA): allowed a significant advance in the personalized management of cancers, as a non-invasive test capable of producing diagnostic, prognostic, theranostic, and of therapeutic follow-up type. The teams of the IRCM of Montpellier have developed a test called IntPlex®, capable of allowing the multiparametric analysis of this cfDNA.

This innovative technology has been patented and validated technically and clinically on large cohorts of patients with different types of cancer and for several types of genetic mutations. Briefly, this Intplex® technology enables the simultaneous determination of five cfDNA measurement and characterization parameters: total cfDNA concentration, fragmentation, point mutation detection, mutant cfDNA concentration and mutational load.

Plasma cfDNA concentrations in patients with CRC are significantly higher than in healthy individuals. These concentrations decrease progressively in patients in remission while they increase in the patients evolutionary or in recurrence. This measure also proves to be an excellent tool to discriminate patients with metastatic CRC from those with more pejorative prognosis. The aim of the work is to measure the cfDNA concentration in subjects undergoing colonoscopy because of a positive immunological fecal test.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ at 18 years old,
* Patient with a positive immunological screening test,
* Patient requiring a colonoscopy
* Patient having given his informed, written and express consent.

Exclusion Criteria:

* Patient not affiliated to a social security scheme,
* Subject under tutelage, curatorship or safeguard of justice,
* Patient in an emergency situation,
* Acute or chronic inflammatory disease,
* Patient having made an intense effort 3 days before sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
AUC | Until the study completion of 2 years
  Area under the ROC curve (AUC) of the total cfDNA concentration.

SECONDARY OUTCOMES:
cfDNA threshold | Until the study completion of 2 years
  Optimal threshold of CfDNA (according to Youden Index)
Intplex parameters | Until the study completion of 2 years
  Sensitivity, specificity, positive predictive value, negative predictive value of the test Intplex

CONTACTS AND LOCATIONS:
Overall Officials: ADENIS Antoine, MD, Study Chair — Institut régional du Cancer de Montpellier
Locations (1):
- ICM - Institut régional du Cancer Montpellier, Montpellier, Occ, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Segnan N, Armaroli P, Bonelli L, Risio M, Sciallero S, Zappa M, Andreoni B, Arrigoni A, Bisanti L, Casella C, Crosta C, Falcini F, Ferrero F, Giacomin A, Giuliani O, Santarelli A, Visioli CB, Zanetti R, Atkin WS, Senore C; SCORE Working Group. Once-only sigmoidoscopy in colorectal cancer screening: follow-up findings of the Italian Randomized Controlled Trial--SCORE. J Natl Cancer Inst. 2011 Sep 7;103(17):1310-22. doi: 10.1093/jnci/djr284. Epub 2011 Aug 18. PMID 21852264
- [Result] Schoen RE, Pinsky PF, Weissfeld JL, Yokochi LA, Church T, Laiyemo AO, Bresalier R, Andriole GL, Buys SS, Crawford ED, Fouad MN, Isaacs C, Johnson CC, Reding DJ, O'Brien B, Carrick DM, Wright P, Riley TL, Purdue MP, Izmirlian G, Kramer BS, Miller AB, Gohagan JK, Prorok PC, Berg CD; PLCO Project Team. Colorectal-cancer incidence and mortality with screening flexible sigmoidoscopy. N Engl J Med. 2012 Jun 21;366(25):2345-57. doi: 10.1056/NEJMoa1114635. Epub 2012 May 21. PMID 22612596
- [Result] Minozzi S, Armaroli P, Segnan N. European guidelines for quality assurance in colorectal cancer screening and diagnosis. First Edition--Principles of evidence assessment and methods for reaching recommendations. Endoscopy. 2012 Sep;44 Suppl 3:SE9-14. doi: 10.1055/s-0032-1309781. Epub 2012 Sep 25. PMID 23012125
- [Result] US Preventive Services Task Force; Bibbins-Domingo K, Grossman DC, Curry SJ, Davidson KW, Epling JW Jr, Garcia FAR, Gillman MW, Harper DM, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Owens DK, Phillips WR, Phipps MG, Pignone MP, Siu AL. Screening for Colorectal Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2016 Jun 21;315(23):2564-2575. doi: 10.1001/jama.2016.5989. PMID 27304597
- [Result] Mouliere F, El Messaoudi S, Pang D, Dritschilo A, Thierry AR. Multi-marker analysis of circulating cell-free DNA toward personalized medicine for colorectal cancer. Mol Oncol. 2014 Jul;8(5):927-41. doi: 10.1016/j.molonc.2014.02.005. Epub 2014 Mar 24. PMID 24698732